CLINICAL TRIAL: NCT07271108
Title: The Effect of Carrying Heavy Shopping Bags on Muscle Function and Mass: a Randomized Controlled Trial.
Brief Title: Carrying Heavy Shopping Bags and Muscle Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Stuart Gray, Prof. of Muscle and Metabolic Health, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200220195
Record Dates: First submitted 2025-11-17; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Strength; Strength Training Effects; Resistance Exercise
Keywords: Health promotion; Resistance training; strength training; carrying shopping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Usual routine (No Intervention)
- Shopping bag carrying (Experimental): Four-week shopping bag carry intervention (15 mins, 2x per week). Performed under supervision in laboratory.
  Interventions: Behavioral: Experimental: Shopping bag carrying

INTERVENTIONS:
Behavioral: Experimental: Shopping bag carrying — Four-week shopping bag carry intervention (15 mins, 2x per week). Performed under supervision in laboratory.
  Arms: Shopping bag carrying

SUMMARY:
What Is This Study About? To find out whether carrying heavy shopping bags twice a week can help adults not currently meeting physical activity strength guidelines improve muscle mass, strength, power, and endurance.

What Can Be learnt?

* Can carrying shopping bags help improve muscle mass, strength, power, and endurance?
* Should carrying shopping bags be included within physical activity recommendations?

Two groups will be compared:

* One group will carry shopping bags twice a week within a controlled lab environment
* The other group won't change anything in their routine.

What Will Participants Do?

* Self-select a weight for shopping bags that is heavy but can be carried for 15 minutes to use for all sessions
* Walk with shopping bags for 15 minutes at a normal walking speed for carrying shopping home from the supermarket.
* After each minute, the time stops and participants place bags on the floor. The time restarts for the next minute when the participant chooses to pick up the bags again.

ELIGIBILITY:
Inclusion Criteria:

* Performing less than 2 days per week of muscle strengthening exercise
* Pass the physical activity readiness questionnaire
* Available during data collection period

Exclusion Criteria:

* Current or prior history of heart, lung, kidney, endocrine or liver disease or cancer.
* Performing more than 2 days per week of muscle strengthening exercise
* Answered yes to any of the questions in the Physical Activity Readiness Questionnaire
* Available during data collection period

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Back strength | Baseline and one week after the intervention ended
  Takei Back Strength Dynamometer (T.K.K. 5002 BACK-A Type-3) used to measure back strength to the nearest 1 kg. Measurements taken with the legs, back and arms straight and the torso flexed to 30 degrees at the hip with the handle held in a natural grip. Participants instructed to gradually pull as hard as they could on the handle in order to raise the upper part of their body without bending their knees. Three trials performed with the maximum value used in the analysis.
Jump Height | Baseline and one week after the intervention ended
  Assessed using a countermovement jump with hands on hips. Participants instructed to crouch into a squat position and then jump as high as possible with legs fully extended and landing on the same spot with knees extended and feet together. After a familiarisation attempt, participants to perform three countermovement jumps and the maximum peak power used in the analysis. Jump height and flight time calculated using Microgate Optojump Next software version 1.10.5.0 connected to photoelectric bars RX10 and TX10 (Microgate Optojump Next, Bolzano, Italy) placed parallel to each other.
  Jump height derived from the equation: H = g×t2/8 (H = the jump height (m), t = jump flight time (seconds) and g = acceleration due to gravity (9.81 m/s-2))
Peak Power | Baseline and one week after the intervention ended
  Assessed using a countermovement jump with hands on hips. Participants instructed to crouch into a squat position and then jump as high as possible with legs fully extended and landing on the same spot with knees extended and feet together. After a familiarisation attempt, participants to perform three countermovement jumps and the maximum peak power used in the analysis. Jump height and flight time calculated using Microgate Optojump Next software version 1.10.5.0 connected to photoelectric bars RX10 and TX10 (Microgate Optojump Next, Bolzano, Italy) placed parallel to each other.
  Peak Power calculated using the Sayers equation: Peak Power (Watts) = 60.7 × jump height (cm) + 45.3 × body mass (kg) - 2055
Muscle Endurance | Baseline and one week after the intervention ended
  Endurance assessed by a 60 second sit to stand test using a 46.5cm high, straight-backed chair with a hard seat and no arm rests. From a seated position with hands on shoulders and arms crossed across the chest, participants instructed to stand up from the chair until their legs were completely straight, then sit back down again (one complete sit to stand) as many times as possible in 60 seconds. The number of complete sit to stands used in the analysis.
Grip strength | Baseline and one week after the intervention ended
  Jamar hydraulic hand dynamometer in handle position II used to measure grip strength to the nearest 1 kg. Measurements taken with the participant seated with feet flat on the floor, elbow flexed 90 degrees by their side and with the wrist just over the end of the arm of the chair in a neutral position (thumbs-up position). Participants instructed to squeeze as hard as possible until the needle stopped rising with the verbal encouragement of "squeeze, squeeze, squeeze and relax". Three trials performed on each side, alternately, with the maximum value used in the analysis in accordance with the Southampton protocol
Body composition | Baseline and one week after the intervention ended
  Assessed using a Body Composition Analyzer Type BC-418 MA (Tanita Corporation, Tokyo, Japan) to determine whole body bioimpedance between the hands and feet by applying a constant current of 90 microamps at 50kHz through the body. Measurements taken in the standing position with bare feet placed on the footplate electrodes and the hand grip electrodes held by the side of the body. Whole body impedance used to derive skeletal muscle mass.

SECONDARY OUTCOMES:
Distance shopping carried | 2 x per week at every visit throughout the 4 week intervention
  The number of complete corridor lengths walked with the shopping bags in 15 minutes was recorded for those in the intervention group.
Perceived exertion | 2 x per week at every visit throughout the 4 week intervention
  Perceived exertion was measured using the Borg Rating of Perceived Exertion scale (RPE) [44] from 6-20, with 20 meaning the harderst exertion and 6 the least exertion at the end of each 15-minute carry for those in the intervention group.

CONTACTS AND LOCATIONS:
Locations (1):
- university of glasgow, James Black Building Lab, Glasgow, Glasgow City, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised participant data will be made available by the author upon request. Data and study protocol will be made available as part of publication.